CLINICAL TRIAL: NCT04465578
Title: Incidence of Short-term Urinary Retention After Fascial Retropubic Sling: Prospective and Randomized Analysis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020-0001
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Stress Urinary Incontinence; Urinary Retention Postoperative; Urinary Retention After Procedure
Keywords: Stress urinary incontinence; Pubovaginal sling; Urinary retention
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling tension adjustment by classic technique (Active Comparator): We will adjust the tension of the sling by using the classic technique (2 fingers between the fascia and the knot)
  Interventions: Procedure: Sling tension adjustment by classic technique
- Sling tension adjustment by height of 4 cm (Active Comparator): We will adjust the tension of the sling by using the height between the fascia and the knot of 4cm
  Interventions: Procedure: Sling tension adjustment by height of 4 cm

INTERVENTIONS:
Procedure: Sling tension adjustment by classic technique — We will adjust the tension of the sling by using the classic technique (2 fingers between the fascia and the knot)
  Arms: Sling tension adjustment by classic technique
Procedure: Sling tension adjustment by height of 4 cm — We will adjust the tension of the sling by using the height between the fascia and the knot of 4cm
  Arms: Sling tension adjustment by height of 4 cm

SUMMARY:
The aim of this study is to evaluate the incidence of short-term urinary retention and the cure rate in patients with stress urinary incontinence undergoing surgical treatment with fascial pubovaginal sling with two tension adjustment techniques: the classic adjustment technique ("2 fingers") and measuring the distance between the fixation knot and the aponeurosis of 4 cm.

DETAILED DESCRIPTION:
A randomized double-blind clinical trial will be conducted in women over 18 years of age with stress urinary incontinence and indication for surgical treatment, who have not undergone previous surgical treatment. Postoperative follow-up will be 1 month when the incidence of urinary retention and the rate of cure after the procedure will be evaluated. The incidence of urinary retention in 1 month postoperatively will be evaluated in the two different techniques (post-voiding residue > 200ml or the need for intermittent bladder catheterization) and the cure rate for urinary incontinence (cough test and response "No" to the question 3 of the Urogenital Distress Inventory questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and no improvement with conservative management

Exclusion Criteria:

* Prior anti incontinence surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of urinary retention in short-term after fascial pubovaginal sling | 1 month
  Urinary retention will be considered the need for bladder catheterization or post-voiding residue> 200ml after 1 month), in patients with tension adjustment by the classic technique x node height to the abdominal rectus fascia of 4cm.

SECONDARY OUTCOMES:
To evaluate the incidence of curing stress urinary incontinence in short-term after fascial pubovaginal sling in both groups. | 1 month
  Cure will be considered the answer "NO" to the 3rd question of Urogenital Distress Inventory and a negative cough test.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Rosito, Doctor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No